CLINICAL TRIAL: NCT06672562
Title: A Randomized Pilot Basket Trial of Discovering Our Best Selves: Narrative Enhancement and Cognitive Therapy for Self-stigma Among Youth
Brief Title: Narrative Enhancement and Cognitive Therapy for Self-Stigma in Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 062/2024
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Bipolar Disorder; Multiple Mental Health Conditions
Keywords: stigma; narrative enhancement and cognitive therapy; youth; comorbidity; self-stigma; mental health disorder
MeSH Terms: conditions — Bipolar Disorder; Social Stigma; Mental Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Masking Description: Data analysts will be masked as to treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NECT-Y (Experimental): Virtual 14-week Narrative Enhancement and Cognitive Therapy group intervention that will be co-facilitated by a clinician and peer support worker.
  Interventions: Behavioral: Narrative Enhancement and Cognitive Therapy
- Treatment as usual (Placebo Comparator): No study-specific care will be provided to these participants.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Narrative Enhancement and Cognitive Therapy — NECT-Y consists of 14 90-minute sessions over the course of 14 weeks. The intervention combines psychoeducation, cognitive therapy, narrative therapy, goal-setting and peer support. Each group meeting includes educational materials, reflections, and active exercises that participants are guided through to personalize the content to their experiences. Participants will be provided with a workbook which allows them to follow the activities easier.
  Arms: NECT-Y
Other: Usual care — Standard usual care. No study-specific care, but participants will be provided with information on community resources and support, and will also be encouraged to speak to their clinician if they are interested in learning about other services.
  Arms: Treatment as usual

SUMMARY:
The goal of this pilot clinical trial is to assess the feasibility of conducting a full-scale study to learn if a new youth-adapted Narrative Enhancement and Cognitive Therapy (NECT-Y) reduces self-stigma in youth living with bipolar disorder or multiple mental health conditions. The main questions it aims to answer are:

* What is the feasibility of conducting a definitive clinical trial in terms of recruitment success, study retention/compliance, treatment retention/compliance, and absence of serious adverse events?
* Can facilitators deliver the adapted NECT-Y intervention with fidelity?
* What is the acceptability of the newly adapted NECT-Y intervention among youth participants and facilitators?

Researchers will compare NECT-Y to treatment as usual (TAU).

Participants will take part in a virtual 14-week NECT-Y group intervention or receive TAU. They will also complete questionnaires at three time points (baseline, post-treatment, and follow-up).

DETAILED DESCRIPTION:
The goal of this pilot basket randomized controlled trial (RCT) is to assess the feasibility of conducting a full-scale study to learn if a youth-adapted Narrative Enhancement and Cognitive Therapy (NECT-Y) can reduce self-stigma in youth diagnosed with bipolar disorder (BD) or with multiple mental health conditions (MMHC). More specifically, this trial has three objectives: 1) to assess whether it is feasible to run a definitive RCT of the new NECT-Y intervention, 2) to explore the facilitators' ability to deliver the new intervention with fidelity, and 3) to assess whether the newly adapted version is acceptable to participants and facilitators, including barriers/facilitators to using NECT-Y.

This parallel-arm pilot basket RCT will be conducted to compare NECT-Y to Treatment as Usual (TAU). The two-arm, pilot RCT will be conducted as two samples within a single basket trial and will include 48 participants with BD and 48 participants with MMHC for a total of approx. 96 participants. Participants will be 1:1 randomized to receive NECT-Y (n=48) or TAU (n=48). Five facilitators, including peer co-facilitators, have been recruited and trained to deliver the intervention.

Participants with BD will be recruited from a clinical pool from outpatient hospital clinics in Toronto (CAMH) and London (LHSC), Ontario, as well as from other CAMH studies if they have provided consent to be re-contacted. Participants with MMHC will be recruited from CAMH only, from among participants recruited to other studies and who have consented to be contacted about additional research opportunities. All participants will follow the same study design. Participants will be screened sequentially during the recruitment period, until the sample size is reached. Eligible participants will complete baseline assessments and then be subsequently randomized to NECT-Y for 14 weeks or TAU. The NECT-Y intervention will be delivered virtually to ≈12 participants/group, with the same number of control participants assigned to TAU. TAU participants will be provided with information on community resources and support, and will also be encouraged to speak to their clinician if they are interested in learning about other services. No study-specific care will be provided to TAU participants. NECT-Y and TAU participants will complete post-treatment assessments after 14 weeks, and again at 3 months follow up. To understand the acceptability of the intervention, qualitative focus groups (approx. 2 hours) will be conducted by the research staff with NECT-Y participants (who consent), and individual interviews will be conducted with the NECT-Y facilitators and peer co-facilitators. Participants randomized to TAU will not receive NECT-Y after the 14-week period as this is beyond the scope of this pilot trial.

This is a youth-engaged mixed methods pilot acceptability and feasibility RCT, with the qualitative component embedded at the post-treatment follow-up stage. Evaluation will include baseline, post-treatment, and 3-month follow-up, feasibility metrics, interpreted together with the themes generated from qualitative focus groups/interviews conducted with participants and facilitators. Lived experience team members will be involved in all stages, from study design to knowledge translation, as co-investigators and a youth advisory group.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of bipolar disorder (any subtype) OR diagnosed with multiple mental health conditions (excluding bipolar disorder)
* 'Mild' to 'severe' internalized stigma (mean score > 2.0 on the Internalized Stigma of Mental Illness Inventory)
* Must sign and date the informed consent form
* Stated willingness to comply with all study procedures

Exclusion Criteria:

* Mental health-related hospitalization or emergency department visit in the last 30 days
* Initiation of a new psychotherapy in the last 30 days
* Inability to consent or to communicate in English

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Providing Consent to Participate in the Study | Duration of the study enrollment period, up to 1 year
  Our study target is > 60% of individuals approached/contacted will consent to participate in the study.
Number of Participants Providing Consent in Two Months | Duration of the study enrollment period, up to 1 year
  The study target is to obtain study consent from 24 participants in two months.
Number of Sessions Attended by Participants Randomized to NECT-Y | From week 1 to week 14 of the NECT-Y intervention, up to 14 weeks
  The study target is that participants randomized to NECT-Y attend > 80% of the 14 sessions.
Number of Participants Completing Study Questionnaires at Week 15 | Week 15 (post-treatment)
  The study target is > 80% of the participants complete at least one questionnaire at post-treatment (week 15).
Number of Participants Completing Study Questionnaires at Week 28 | Week 28 (3-month follow up)
  The study target is > 80% of the participants complete at least one questionnaire at 3-month follow up (week 28).
Number of Questionnaires Completed at Week 15 | Week 15 (post-treatment)
  The study target is participants complete > 90% of the 14 questionnaires at post-treatment (week 15).
Number of Questionnaires Completed at Week 28 | Week 28 (3-month follow up)
  The study target is participants complete > 90% of the 14 questionnaires at 3-month follow up (week 28).
Number of Participants With Study-Related Adverse Events as Assessed by an Institutional Adverse Event Log | From study enrollment to 3-month follow up, up to 28 weeks
  The study target is for their to be no adverse events throughout a participants enrollment in the study, including no AEs from participating in the NECT-Y intervention. AEs will be tracked ad hoc as participants self-report any AEs.

SECONDARY OUTCOMES:
Was NECT-Y Acceptable to Youth Participants? | ~ Week 15 (2-hour focus group)
  Qualitative measure assessed in focus groups. Individuals will be asked to comment on their experience receiving NECT-Y, their impressions of the youth adaptation, and whether it was an appropriate intervention.
Was NECT-Y Acceptable to Co-Facilitators? | ~ Week 28 (1-hour interview)
  Qualitative measure assessed in qualitative interviews. Individuals will be asked to comment on their experience facilitating NECT-Y, their impressions of the youth adaptation, and whether it was an appropriate intervention.
Was NECT-Y Delivered With Fidelity in Relation to the Intervention Manual as Assessed by a Standardized Fidelity Scale? | From week 1 to week 14 of the NECT-Y intervention, up to 14 weeks
  Scale: NECT Fidelity Scale; 8-item scale, minimum value 1 (Poor), maximum value 5 (Excellent). Higher scores indicate greater fidelity in how the group facilitators delivered NECT-Y as intended based on the intervention manual. Conducted for each NECT-Y group. Sessions will be audio-recorded and rated. Two trained staff will code the recordings, and inter-rated reliability will be calculated and fidelity scores computed. Target is a mean overall fidelity rating of 4 on a 5-point scale.

OTHER OUTCOMES:
Change from Baseline in the Mean Self-Stigma at Week 15 (post-treatment) | baseline, 15 weeks
  Scale: Internalized Stigma of Mental Illness Inventory; 29 item scale, minimum value for each item = 0 (Strongly disagree), maximum value = 3 (Strongly agree). Higher scores indicate more severe self-stigma.
Change from Baseline in the Mean Self-Stigma at Week 28 (3-Months Follow-up) | baseline, 28 weeks
  Scale: Internalized Stigma of Mental Illness Inventory; minimum value for each item = 0 (Strongly disagree), maximum value = 3 (Strongly agree). Higher scores indicate more severe self-stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hawke, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data will be placed in a local brain health data bank following institutional requirements.

REFERENCES:
- [Background] Hawke LD, Bennett R, Sheikhan NY, Yanos P. Lived experience adaptation of a psychosocial intervention for young adults with bipolar spectrum disorders: Process description and adaptation outcomes. Early Interv Psychiatry. 2023 Nov;17(11):1125-1130. doi: 10.1111/eip.13461. Epub 2023 Aug 31. PMID 37650493
- [Derived] Hawke LD, Husain MI, Amartey A, Ma C, Osuch E, Yanos PT, Gallagher L, Jordan A, Orson J, Lee A, Kozloff N, Kidd SA, Goldstein BI, Sheikhan NY, Ortiz A, Szatmari P. Narrative enhancement and cognitive therapy for self-stigma among youth with bipolar disorder or multiple mental health conditions: protocol for a pilot randomised basket trial. BMJ Open. 2025 Feb 26;15(2):e096222. doi: 10.1136/bmjopen-2024-096222. PMID 40010812